CLINICAL TRIAL: NCT02868736
Title: Clinical Validation of CD Diagnostics Synovasure PJI ELISA Test and Synovasure PJI Lateral Flow Test for Detection of Periprosthetic Joint Infection in Synovial Fluid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CD Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CDD-CLI-001
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Periprosthetic Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected Periprosthetic Joint Infection: Individuals who are suspected of having Periprosthetic Joint Infection (PJI)
  Interventions: Device: Synovasure PJI Lateral Flow test and Synovasure PJI ELISA Test

INTERVENTIONS:
Device: Synovasure PJI Lateral Flow test and Synovasure PJI ELISA Test

SUMMARY:
* To demonstrate the tests' performance when compared to the detection of PJI using the Musculoskeletal Infection Society (MSIS) criteria-based definition of PJI for diagnosing PJI.1 This criteria-based definition of PJI places emphasis on culture techniques that identify pathogens, but also provides for minor criteria that can be used to diagnose PJI;
* To calculate the tests' clinical sensitivity, clinical specificity, positive predictive value (PPV), and negative predictive value (NPV).

DETAILED DESCRIPTION:
A major disadvantage of the MSIS criteria-based definition of PJI is that two of the essential criteria, tissue culture and histological analysis, are only available after surgery. In cases where the surgical samples are critical for the diagnosis of infection, the physician may need to adjust his or her treatment post operatively for the patient based on the treatment provided. The availability of a preoperative test that correlates well with the MSIS criteria could improve patient care. Currently, when a clinician is suspicious of PJI due to pain or failure of an arthroplasty, it is considered the standard-of-care to request blood and synovial fluid tests to begin the process of diagnosing infection. A synovial fluid test for PJI that correlates with the final MSIS definition could be requested at this early preoperative stage of the diagnostic process.

Synovasure® PJI ELISA Test is a qualitative in vitro diagnostic device intended as an adjunct for the detection of periprosthetic joint infection (PJI) in synovial fluid from patients being evaluated for revision surgery. Synovasure® PJI ELISA Test utilizes a test that measures biomarkers, alpha-defensins 1-3, in the synovial fluid of joints that are infected. Synovasure® PJI ELISA Test results are intended to be used in conjunction with other clinical and diagnostic findings to aid in a patient's diagnosis of infection.

Synovasure® PJI Lateral Flow Test is a qualitative in vitro diagnostic device intended as an adjunct for the detection of periprosthetic joint infection (PJI) in synovial fluid from patients being evaluated for revision surgery. Synovasure® PJI Lateral Flow Test utilizes a test that measures biomarkers, alpha-defensins 1-3, in the synovial fluid of joints that are infected. Synovasure® PJI Lateral Flow Test results are intended to be used in conjunction with other clinical and diagnostic findings to aid in a patient's diagnosis of infection.

ELIGIBILITY:
Inclusion Criteria:

* • Subject has a total knee and/or hip joint arthroplasty.

  * The subject will be evaluated for revision surgery.

    o Operative samples are required for full MSIS classification.
  * Subject is ≥22 years of age.
  * Subject has had no recent injections or surgeries of the joint (within past 6 weeks).
  * Subject has or will have all of the medical tests required to allow MSIS classification.
  * Subject signs informed consent form.

Exclusion Criteria:

* • Subject does not have a total knee and/or hip joint arthroplasty.

  * Healthy subjects without medical need for aspiration.
  * Subject did not have a revision surgery.
  * Subjects with a diagnostic synovial fluid specimen collection within the past 14 days.
  * Subjects <22 years of age.
  * Subject has had an injection, lavage, or surgery of the joint within the past 6 weeks.
  * Subject does not have all of the medical tests required for MSIS classification.
  * Subject does not sign informed consent form.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a total knee and/or hip joint replacement and are being evaluated for revision surgery will be recruited for the trial.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of laboratory results and physical findings required to diagnose PJI | Outcome is measured at time of aspiration and again at time of revision surgery.
  The clinical endpoint for the study is Adjudication Panel evaluation of the laboratory results and physical findings required to diagnose PJI. There are two major criteria, and five minor criteria in the MSIS definition of PJI. The existence of one positive major criterion is sufficient for the diagnosis of PJI. Similarly, the existence of any three of the five positive minor criteria is considered sufficient for the diagnosis of PJI.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States